CLINICAL TRIAL: NCT05592691
Title: Ropivacaine Plasma Concentrations After Fascial Blocks in Elective Cardio-thoracic and Abdominal Surgery: an Observational, Monocentric Study
Brief Title: Ropivacaine Plasma Concentrations After Fascial Blocks in Elective Cardio-thoracic and Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Luca Brazzi, Full Professor, Director, University of Turin, Italy
Other Study IDs: PRAST
Record Dates: First submitted 2022-09-21; First posted 2022-10-25 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Local Anesthetic Toxicity; Regional Anesthesia Morbidity; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: Patients undergoing fascial blocks in elective cardio-thoracic and abdominal surgery.
  Interventions: Procedure: Fascial block

INTERVENTIONS:
Procedure: Fascial block — The end of the drug infusion will be considered the time zero (T0); subsequently blood samples (4ml) will be taken at pre-established time intervals (after 5, 15, 30, 60, 120 and 180 minutes). Blood samples will be collected in test tubes and centrifuged within 1 hour of collection; subsequently they will be stored at a low temperature and transported to the reference analysis laboratory.

SUMMARY:
Primary aim: observe the incidence of systemic toxicity from local anesthetic (LAST) after performing fascial blocks in patients undergoing elective cardio-thoracic and abdominal surgery.

Secondary aim: describe the pharmacokinetic profile of the local anesthetic (ropivacaine) and assess peri-procedural complications, post-operative pain and opiate consumption in the first 24 hours.

DETAILED DESCRIPTION:
Loco-regional anesthesia (LRA) procedures have acquired, in recent years, increasing importance in the peri-operative control of pain in the field of cardio-thoracic and abdominal surgery. To date, they are recognized as part of the multimodal analgesia underlying the Enhanced Recovery After Surgery (ERAS) protocols as they have demonstrated a better efficacy in post-operative pain control than the use of opiates alone and allow a significant reduction in the use of opioids in the postoperative period.

The advent of ultrasound-guided LRA procedures has led to the development of numerous fascial blocks, which involve the injection, at the level of the muscle-fascial planes, of an abundant volume of low-concentration local anesthetic to allow spread to adjacent nerve structures. The fascial blocks represent a valid alternative to epidural analgesia for the control of postoperative pain in the thoracoabdominal area, as they are characterized by a rapid learning curve and a lower risk of periprocedural complications compared to neuraxial anesthesia procedures.

The main chest wall nerve blocks used in clinical practice include the pectoral nerve block (PECS1 and PECS2) and serrate anterior plane block (SAP) at the level of the anterior chest wall; the spinal erector plane (ESP) block and the paravertebral block at the level of the posterior thoracic wall.

LRA techniques also play a fundamental role in the field of abdominal surgery, especially in the context of multimodal analgesia, aiming to reduce consumption and, consequently, the secondary side effects of the use of opioids.

In the case of laparotomic major abdominal surgery, the use of epidural analgesia has been shown to be effective in reducing post-operative pain, opioid consumption, and recovery of gastrointestinal function, but has not shown a significant reduction in the duration of hospitalization and of post-operative complications.

Subarachnoid analgesia is mainly indicated in laparoscopic abdominal surgery. Numerous studies have shown an efficacy similar to epidural anesthesia in controlling pain and reducing opioid consumption as well as allowing early patient mobilization and a shorter length of hospital stay.

The transverse abdominal plane (TAP) block has a rapid learning curve and has been shown to be effective in controlling postoperative analgesia, reducing opioids consumption and reducing hospital stay.

The lumbar square (QoL) block has a greater efficacy than other abdominal wall blocks on the visceral component of pain. A recent meta-analysis demonstrated greater efficacy than TAP in the control of post-operative pain and guarantees a longer duration of analgesia.

The effectiveness of the anesthetic depends on its local action at the level of the nervous structures "wetted" by the drug; a variable amount of local anesthetic undergoes systemic absorption and might be responsible for part of the analgesic effect, but above all for the possible appearance of systemic side effects.10 The amount of drug redistributing in the blood depends on the total dose of the drug administered, the route of administration, and the vascularity of the injection site.

Ropivacaine is a long-acting amide local anesthetic frequently used in LRA procedures. Unlike other drugs of the same family, the levorotatory enantiomer S-Ropivacaine is characterized by reduced lipophilicity and this determines a lower risk of toxicity to the Central Nervous System (CNS) and cardiovascular system (CVS). The drug exhibits high plasma protein binding (α1-acid glycoprotein), linear absorption kinetics, hepatic metabolism, and renal elimination.

Systemic toxicity from Local anesthetic (LAST) represents a complication of local anesthetic administration and is directly dependent on the plasma concentration of the drug. The signs and symptoms of LAST occur progressively and mainly affect the CNS (visual disturbances, perioral hypoaesthesia, dizziness, euphoria, muscle stiffness, spasms, convulsions) and the CVS system (hypotension, bradycardia, arrhythmias, cardiac arrest).

The study aims to observe the onset of local anesthetic toxicity (LAST) after performing fascial blocks in patients undergoing elective cardiothoracic and abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardio-thoracic and abdominal surgery with indications for the execution of fascial block
* Signature of the informed consent form.

Exclusion Criteria:

* Lack of informed consent form.
* Previous neuropsychiatric pathologies or neuropathies of the back / trunk
* Severe renal insufficiency (GFR <30ml / min)
* Severe hepatic insufficiency or alteration of liver enzymes
* Contraindications to LRA procedures (injection site infection, coagulopathy, allergy / hypersensitivity to local anesthetics)
* Pregnancy
* Hypoalbuminemia
* Hospitalization in intensive care and / or post-operative sedation> 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the enrollment of patients who will undergo elective cardio-thoracic and / or abdominal surgery at the A.O.U. Città della Salute e della Scienza of Turin, with clinical indications for the execution of band blocks for analgesic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of systemic toxicity from local anesthetic signs and symptoms. | 6 hours after surgery
  The typical presentation of LAST usually begins with prodromal symptoms and signs, such as perioral numbness, tinnitus, agitation, dysarthria, and confusion. These may be followed by more severe central nervous system (CNS) derangements such as seizures and coma.
Incidence of systemic toxicity from local anesthetic signs and symptoms. | 12 hours after surgery
  The typical presentation of LAST usually begins with prodromal symptoms and signs, such as perioral numbness, tinnitus, agitation, dysarthria, and confusion. These may be followed by more severe central nervous system (CNS) derangements such as seizures and coma.
Incidence of systemic toxicity from local anesthetic signs and symptoms. | 24 hours after surgery
  The typical presentation of LAST usually begins with prodromal symptoms and signs, such as perioral numbness, tinnitus, agitation, dysarthria, and confusion. These may be followed by more severe central nervous system (CNS) derangements such as seizures and coma.

SECONDARY OUTCOMES:
Ropivacaine concentration | 5 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine concentration | 15 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine concentration | 30 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine concentration | 60 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine concentration | 120 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine concentration | 180 minutes from the fascial block execution
  Ropivacaine plasma concentration
Ropivacaine latency time | 5 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Ropivacaine latency time | 15 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Ropivacaine latency time | 30 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Ropivacaine latency time | 60 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Ropivacaine latency time | 120 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Ropivacaine latency time | 180 minutes from the fascial block execution
  Ropivacaine maximum plasma concentration and latency time between the execution of the block and the achievement of Cmax
Anesthesia effectiveness | Immediately after fascial block
  Global extension of the anesthetized skin surface, measured by Pinprick test.
Post-operative pain | 0 hours after awakening
  Pain after awakening, estimated using the numeric scale for pain assessment (min 0 max 10, 10 equals worst outcome)
Post-operative pain | 1 hour after awakening
  Pain after awakening, estimated using the numeric scale for pain assessment (min 0 max 10, 10 equals worst outcome)
Post-operative pain | 6 hours after awakening
  Pain after awakening, estimated using the numeric scale for pain assessment (min 0 max 10, 10 equals worst outcome)
Post-operative pain | 12 hours after awakening
  Pain after awakening, estimated using the numeric scale for pain assessment (min 0 max 10, 10 equals worst outcome)
Post-operative pain | 24 hours after awakening
  Pain after awakening, estimated using the numeric scale for pain assessment (min 0 max 10, 10 equals worst outcome)
Opioid requirement | 0 hours after awakening
  Pain after awakening, estimated using morphine equivalent milligrams
Opioid requirement | 1 hour after awakening
  Pain after awakening, estimated using morphine equivalent milligrams
Opioid requirement | 6 hours after awakening
  Pain after awakening, estimated using morphine equivalent milligrams
Opioid requirement | 12 hours after awakening
  Pain after awakening, estimated using morphine equivalent milligrams
Opioid requirement | 24 hours after awakening
  Pain after awakening, estimated using morphine equivalent milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Ceraolo, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Turin, Italy

REFERENCES:
- [Background] Crumley S, Schraag S. The role of local anaesthetic techniques in ERAS protocols for thoracic surgery. J Thorac Dis. 2018 Mar;10(3):1998-2004. doi: 10.21037/jtd.2018.02.48. PMID 29707356
- [Background] Chin KJ, Versyck B, Pawa A. Ultrasound-guided fascial plane blocks of the chest wall: a state-of-the-art review. Anaesthesia. 2021 Jan;76 Suppl 1:110-126. doi: 10.1111/anae.15276. PMID 33426660
- [Background] Jack JM, McLellan E, Versyck B, Englesakis MF, Chin KJ. The role of serratus anterior plane and pectoral nerves blocks in cardiac surgery, thoracic surgery and trauma: a qualitative systematic review. Anaesthesia. 2020 Oct;75(10):1372-1385. doi: 10.1111/anae.15000. Epub 2020 Feb 16. PMID 32062870
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Hughes MJ, Ventham NT, McNally S, Harrison E, Wigmore S. Analgesia after open abdominal surgery in the setting of enhanced recovery surgery: a systematic review and meta-analysis. JAMA Surg. 2014 Dec;149(12):1224-30. doi: 10.1001/jamasurg.2014.210. PMID 25317633
- [Background] Leone S, Di Cianni S, Casati A, Fanelli G. Pharmacology, toxicology, and clinical use of new long acting local anesthetics, ropivacaine and levobupivacaine. Acta Biomed. 2008 Aug;79(2):92-105. PMID 18788503